CLINICAL TRIAL: NCT02412995
Title: The Effects of Sea Buckthorn and Strawberry on Postprandial Glycaemia, Insulinemia and Appetite - A Randomised, Controlled, Crossover Study of Danish Berries in Overweight and Obese Male Subjects
Brief Title: The Effects of Sea Buckthorn and Strawberry on Postprandial Glycaemia, Insulinemia and Appetite
Acronym: OPUS-WP3C
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Nordea-fonden (Unknown)
Responsible Party: Principal Investigator, Professor Lars Ove Dragsted, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: M208
Record Dates: First submitted 2015-02-08; First posted 2015-04-09 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Insulin Sensitivity; Glucose Intolerance
Keywords: sea buckthorn; strawberry; glucose response; satiety; metabolomics; intake biomarker
MeSH Terms: conditions — Insulin Resistance; Glucose Intolerance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Meal sequence 1-2-3 (Experimental): The three meals, sea buckthorn puree, strawberry puree, or placebo (sugar drink) were allocated a number (1-3) in a blinded fashion and given to the participants in the order 1-2-3
  Interventions: Other: Meal sequence 1-2-3
- Meal sequence 1-3-2 (Experimental): The three meals, sea buckthorn puree, strawberry puree, or placebo (sugar drink) were allocated a number (1-3) in a blinded fashion and given to the participants in the order 1-3-2
  Interventions: Other: Meal sequence 1-3-2
- Meal sequence 2-3-1 (Experimental): The three meals, sea buckthorn puree, strawberry puree, or placebo (sugar drink) were allocated a number (1-3) in a blinded fashion and given to the participants in the order 2-3-1
  Interventions: Other: Meal sequence 2-3-1
- Meal sequence 2-1-3 (Experimental): The three meals, sea buckthorn puree, strawberry puree, or placebo (sugar drink) were allocated a number (1-3) in a blinded fashion and given to the participants in the order 2-1-3
  Interventions: Other: Meal sequence 2-1-3
- Meal sequence 3-1-2 (Experimental): The three meals, sea buckthorn puree, strawberry puree, or placebo (sugar drink) were allocated a number (1-3) in a blinded fashion and given to the participants in the order 3-1-2
  Interventions: Other: Meal sequence 3-1-2
- Meal sequence 3-2-1 (Experimental): The three meals, sea buckthorn puree, strawberry puree, or placebo (sugar drink) were allocated a number (1-3) in a blinded fashion and given to the participants in the order 3-2-1
  Interventions: Other: Meal sequence 3-2-1

INTERVENTIONS:
Other: Meal sequence 1-2-3 — The subjects were studied in three 2 h meal tests with a subsequent ad libitum meal on separate days, at least two days apart. The subjects were individually randomised to the sequence of the test meals using random permutation. The study included two berry meals based on 150 g of frozen berries; sea buckthorn (Hippophaë rhamnoides) and strawberry (Fragaria x ananassa), respectively, and one control meal which did not contain berries. Each meal contained 35 g of sucrose and was adjusted for protein and fat with whey protein and canola oil, respectively. The meals were served with 120 mL of water.
  Arms: Meal sequence 1-2-3
Other: Meal sequence 1-3-2 — The subjects were studied in three 2 h meal tests with a subsequent ad libitum meal on separate days, at least two days apart. The subjects were individually randomised to the sequence of the test meals using random permutation. The study included two berry meals based on 150 g of frozen berries; sea buckthorn (Hippophaë rhamnoides) and strawberry (Fragaria x ananassa), respectively, and one control meal which did not contain berries. Each meal contained 35 g of sucrose and was adjusted for protein and fat with whey protein and canola oil, respectively. The meals were served with 120 mL of water.
  Arms: Meal sequence 1-3-2
Other: Meal sequence 2-3-1 — The subjects were studied in three 2 h meal tests with a subsequent ad libitum meal on separate days, at least two days apart. The subjects were individually randomised to the sequence of the test meals using random permutation. The study included two berry meals based on 150 g of frozen berries; sea buckthorn (Hippophaë rhamnoides) and strawberry (Fragaria x ananassa), respectively, and one control meal which did not contain berries. Each meal contained 35 g of sucrose and was adjusted for protein and fat with whey protein and canola oil, respectively. The meals were served with 120 mL of water.
  Arms: Meal sequence 2-3-1
Other: Meal sequence 2-1-3 — The subjects were studied in three 2 h meal tests with a subsequent ad libitum meal on separate days, at least two days apart. The subjects were individually randomised to the sequence of the test meals using random permutation. The study included two berry meals based on 150 g of frozen berries; sea buckthorn (Hippophaë rhamnoides) and strawberry (Fragaria x ananassa), respectively, and one control meal which did not contain berries. Each meal contained 35 g of sucrose and was adjusted for protein and fat with whey protein and canola oil, respectively. The meals were served with 120 mL of water.
  Arms: Meal sequence 2-1-3
Other: Meal sequence 3-1-2 — The subjects were studied in three 2 h meal tests with a subsequent ad libitum meal on separate days, at least two days apart. The subjects were individually randomised to the sequence of the test meals using random permutation. The study included two berry meals based on 150 g of frozen berries; sea buckthorn (Hippophaë rhamnoides) and strawberry (Fragaria x ananassa), respectively, and one control meal which did not contain berries. Each meal contained 35 g of sucrose and was adjusted for protein and fat with whey protein and canola oil, respectively. The meals were served with 120 mL of water.
  Arms: Meal sequence 3-1-2
Other: Meal sequence 3-2-1 — The subjects were studied in three 2 h meal tests with a subsequent ad libitum meal on separate days, at least two days apart. The subjects were individually randomised to the sequence of the test meals using random permutation. The study included two berry meals based on 150 g of frozen berries; sea buckthorn (Hippophaë rhamnoides) and strawberry (Fragaria x ananassa), respectively, and one control meal which did not contain berries. Each meal contained 35 g of sucrose and was adjusted for protein and fat with whey protein and canola oil, respectively. The meals were served with 120 mL of water.
  Arms: Meal sequence 3-2-1

SUMMARY:
The effects of strawberry and sea buckthorn on postprandial glycaemia and insulinemia as well as on metabolic profiles were examined in overweight or obese male subjects. The study was conducted as a randomised, controlled, single-blinded, 3-way crossover study. Eighteen subjects were studied in three 2 h meal tests followed by a subsequent ad libitum meal. Test meals contained either sea buckthorn, strawberry or no berries and added sucrose to match with respect to sucrose content. Blood samples were collected at baseline and several times postprandially. Subjective appetite sensations were recorded at baseline and every 15-20 min until 140 min and a subsequent ad libitum intake was recorded. Urine samples were also collected at baseline and at several time intervals until 24 hours. Blood and urine were subjected to metabolic profiling to investigate potential biomarkers of berry intake.

DETAILED DESCRIPTION:
Purpose: Berries and mixed berry products exert acute effects on postprandial glycaemia and insulinemia, but very few berries have been studied, and primarily in normal weight subjects. Sea buckthorn and strawberry are compositionally widely different berries and may likely produce different responses. The effects of strawberry and sea buckthorn on postprandial glycaemia and insulinemia were examined in overweight or obese male subjects. Subjective appetite sensations and ad libitum intake were also examined. Berries may thus improve health in longer studies; however, accurate assessment of berry intake is still problematic. The discovery of objective biomarkers for intake of berries is therefore important in assessing both intake and compliance. The investigators aimed to identify urinary exposure markers of two very different berries, strawberry and sea buckthorn, in humans.

Methods: The study was conducted as a randomised, controlled, single-blinded, 3-way crossover study. Eighteen subjects were studied in three 2 h meal tests followed by a subsequent ad libitum meal. Test meals contained either sea buckthorn, strawberry or no berries and added sucrose to match with respect to sucrose content. Blood samples were collected at t = 0, 30, 45, 60, 90 and 120 min. Subjective appetite sensations were recorded at t = 0, 15, 30, 45, 60, 90, 120 and 140 min and subsequent ad libitum intake was recorded. Statistical differences in all continuous measures were evaluated based on the existence of a meal or a time-meal interaction by repeated measurements analyses or differences in the area under the curve (AUC) for that measure in a linear mixed model. Urine samples were collected on each test day at t=-15min, t=0-1h, t=1-2h, and t=2-24h and were analyzed by untargeted metabolomics. Multivariate analysis was applied to discover markers, followed by molecular fragmentation to ease their chemical identification.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male, aged 20-50 years and body mass index (BMI) 25-35 kg/m2

Exclusion Criteria:

* Any current or chronic clinical conditions
* Chronic/frequent use of medication
* Smoking
* Blood donation
* High level of strenuous physical activity (>10h/week)
* High habitual alcohol consumption (>14 drinks/week)
* Present or previous drug abuse
* Participation in other human intervention studies, and obesity surgery

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-10; Primary Completion 2012-11 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Glycemia Area under the plasma glucose concentration curve, concentration curve. | postprandially 0-120min
  Area under the plasma glucose concentration curve, concentration curve.

SECONDARY OUTCOMES:
Insulin response Area under the plasma insulin concentration curve | postprandially 0-120min
  Area under the plasma insulin concentration curve
Appetite scores (visual analogue scale) | postprandially 0-140min
  Measured on a 100 mm visual analogue scale spanning the sensation from minimum to maximum on the following: hunger, satiety, fullness, perceived prospective food intake, thirst, well-being, and desire for something sweet.
urine metabolic profile | 0-24 hrs
  Urine samples were collected on each test day at t=-15min, t=0-1h, t=1-2h, and t=2-24h and were analyzed by untargeted metabolomics (UPLC-QTOF)
plasma metabolic profile (metabolic profiling by UPLC-QTOF) | 0-120min
  Blood samples were drawn at t = -20 (baseline), 30, 45, 60, 90 and 120 min on each test day and subjected to untargeted metabolic profiling by UPLC-QTOF
Meal perception VAS questionnaire | postprandially at 30min and 140 min
  A VAS questionnaire concerning meal perception with ratings for taste (poor/good), smell (not appetising/appetising), appearance (not appetising/appetising), undertaste (none/much), and overall impression (not appetising/appetising).
Incremental area under the plasma glucose concentration curve | postprandially, 0-30 and 0-60min
  The area under the initial part of the glucose plasma curve from the volunteer has ingested the sugar solution until 60 min later
Glycemic profile (calculated as the time in minutes during which the blood glucose concentration is above baseline concentration divided by the incremental peak value of blood glucose) | 0-120 min
  Gycemic profile((calculated as the time in minutes during which the blood glucose concentration is above baseline concentration divided by the incremental peak value of blood glucose)
Incremental insulin response Incremental area under the plasma insulin concentration curve. | Postprandially 0-30 and 0-60 min
  Incremental area under the plasma insulin concentration curve.

CONTACTS AND LOCATIONS:
Overall Officials: Lars O Dragsted, Ph.D., Principal Investigator — University of Copenhagen
Locations (1):
- Department of Nutrition, Exercise and Sports, University of Copenhagen, Frederiksberg C, Denmark